CLINICAL TRIAL: NCT04705701
Title: Randomized Controlled Trial of Post Cardiac Surgery Outcomes in End Stage Renal Disease Patients Comparing Early Dialysis on the Day of Surgery Versus Standard Care
Brief Title: Comparing Post Cardiac Surgery Outcomes in ESRD Patient's With Early Dialysis Versus Standard Care
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Trial was withdrawn due to Covid-19 pandemic
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: earlydialysis2021
Record Dates: First submitted 2020-12-07; First posted 2021-01-12 (Actual); Last update posted 2022-12-19 (Actual); Status verified 2022-12

CONDITIONS: Respiratory Failure; Shock; Coagulopathy
MeSH Terms: conditions — Respiratory Insufficiency; Shock; Hemostatic Disorders | interventions — Renal Dialysis

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A group participants receive same day post-op dialysis (Experimental): Arm A group participants receive same day post-op dialysis
  Interventions: Procedure: Hemodialysis
- Arm B group participants receive dialysis per standard care (No Intervention): Arm B group participants receive dialysis per standard care

INTERVENTIONS:
Procedure: Hemodialysis — Renal replacement therapy is considered standard of care for end stage renal disease patients for clearing the blood and also helping with volume optimization, has different modalities, in our study we are using intermittent hemodialysis.
  Arms: Arm A group participants receive same day post-op dialysis

SUMMARY:
End-stage renal disease (ESRD) is an important risk factor for coronary and valvular cardiac disease leading to cardiac surgery. with concern for higher post-op complications with volume overload and coagulopathies in this patient' outcomes as mentioned above in patients who receive early post-op dialysis versus hemodialysis on day 1 or thereafter.

ed for mechanical ventilation and rs of clinical course and mortality. Previous studies have demonstrated that presence of ESRD is an independent risk factor for post-operative respiratory failure and mortality in patients undergoing cardiac surgery, partially mediated through volume overload and prolonged mechanical ventilation, as well as coagulopathy attributed to platelet dysfunction and uremia.

Prolonged mechanical ventilation after cardiac surgery has been shown to be associated with higher morbidity and mortality. Fluid overload is a predictor of length of mechanical ventilation and intensive care unit (ICU) stay. Therefore early restoration of volume and electrolyte homeostasis and clearance of uremic toxins should be one of the principal goals in the immediate post operative period in patients with ESRD. However, to the best of our knowledge, the effect of timing of post-operative renal replacement therapy, specifically hemodialysis, on clinical outcomes has not been studied in ESRD patients undergoing cardiac surgery.

Accordingly, we have conducted this study to evaluate the effect of early population affecting their overall hospital course including longer duration of ICU stay, need for mechanical ventilation support and blood products transfusion we are planning to conduct this study and compare the short term hemodialysis treatment after cardiac surgery, on clinical outcomes related to volume overload and coagulopathy (i.e. duration of mechanical ventilation, transfusion requirements, and length of ICU stay) in patients with ESRD

DETAILED DESCRIPTION:
End-stage renal disease (ESRD) is an important risk factor for coronary and valvular cardiac disease leading to cardiac surgery. Both volume overload and coagulopathy in the immediate post-operative period after cardiac surgery are important predictors of clinical course and mortality. Previous studies have demonstrated that presence of ESRD is an independent risk factor for post-operative respiratory failure and mortality in patients undergoing cardiac surgery, partially mediated through volume overload and prolonged mechanical ventilation, as well as coagulopathy attributed to platelet dysfunction and uremia.

Prolonged mechanical ventilation after cardiac surgery has been shown to be associated with higher morbidity and mortality. Fluid overload is a predictor of length of mechanical ventilation and intensive care unit (ICU) stay. Therefore early restoration of volume and electrolyte homeostasis and clearance of uremic toxins should be one of the principal goals in the immediate post operative period in patients with ESRD. However, to the best of our knowledge, the effect of timing of post-operative renal replacement therapy, specifically hemodialysis, on clinical outcomes has not been studied in ESRD patients undergoing cardiac surgery.

Accordingly, we are planning to conduct this study to evaluate the effect of early hemodialysis treatment after cardiac surgery, on clinical outcomes related to volume overload and coagulopathy (i.e. duration of mechanical ventilation, transfusion requirements, and length of ICU stay) in patients with ESRD

ELIGIBILITY:
Inclusion Criteria:

* All post operative cardiac surgery ESRD patients who are not meeting exclusion criteria (mentioned below) would be included in the study

Exclusion Criteria:

* hyperkalemia serum K>5.5, severe acidosis PH < 7.2, clinical evidences of volume

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2021-09-02 (Estimated); Study Completion 2021-09-02 (Estimated)

PRIMARY OUTCOMES:
length of mechanical ventilation | A minimum of 1 day up to 7 days
  the duration of mechanical ventilation related to pulmonary congestion in anuric end stage kidney disease patients affected by early dialysis and fluid overload optimization
intensive care unit (ICU) stay | A minimum of 1 day up to 7 days
  following above, requirement for mechanical ventilation support and pulmonary edema affected by early dialysis helping fluid overload optimization and earlier weaning from ventilator, therefor shorter ICU stay

SECONDARY OUTCOMES:
blood product requirement postoperatively | A minimum of 1 day up to 7 days
  coagulopathy and platelet dysfunction in end stage kidney disease patients being corrected faster with early dialysis

CONTACTS AND LOCATIONS:
Overall Officials: Maria DeVita, MD, Principal Investigator — Lenox Hill Hospital

IPD SHARING:
Plan to Share IPD: No